CLINICAL TRIAL: NCT05206318
Title: Efficacy and Safety of Topical Cysteamine for Postinflammatory Hyperpigmentation: A Randomized Control, Double Blinded-trial
Brief Title: Efficacy and Safety of Topical Cysteamine for Postinflammatory Hyperpigmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Scientis Pharma SA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202101456A3
Record Dates: First submitted 2022-01-23; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Hyperpigmentation; Postinflammatory
Keywords: Cysteamine; Postinflammatory Hyperpigmentation; Randomized control trial; Double blinded
MeSH Terms: conditions — Hyperpigmentation | interventions — Cysteamine

STUDY DESIGN:
Intervention Model Description: Randomized control trial, Double masked, double-blinded
Who Masked: Participant, Investigator
Masking Description: The packaging and labeling of the topical product were the same in both group. The subjects were randomized in by an interactive web response system that provided study kit number from the randomization list at the time of inclusion into the study. The randomization list was kept strictly confidential throughout the study and was not available to the investigator and patient or any other personnel who may influence the study data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 participants with topical cysteamine cream (Experimental): Participants with post-inflammatory hyperpigmentation will apply topical cysteamine cream for a 16 weeks period.
  Interventions: Drug: Topical Cysteamine
- 20 participants with topical vehicle control cream (Sham Comparator): Participants with post-inflammatory hyperpigmentation will apply topical vehicle-control cream for a 16 weeks period.
  Interventions: Drug: Topical Vehicle Control

INTERVENTIONS:
Drug: Topical Cysteamine — Topical cysteamine cream applied to the postinflammatory hyperpigmentation dark spots 15 minutes per day, followed by a face wash and moisturizing cream.
  Other Names: Cyspera
  Arms: 20 participants with topical cysteamine cream
Drug: Topical Vehicle Control — Topical vehicle control cream without cysteamine active ingredients applied to the postinflammatory hyperpigmentation dark spots 15 minutes per day, followed by a face wash and moisturizing cream.
  Arms: 20 participants with topical vehicle control cream

SUMMARY:
Post-inflammatory hyperpigmentation is a common pigmentary skin disorder that is refractory to treatment. The treatment for postinflammatory hyperpigmentation is limited. Recent studies have shown that the topical skin care product cysteamine cream has a significant decrease in melanin index without obvious side effects in other dark spots such as melasma. The goal of this study is to determine the safety and efficacy of topical cysteamine in the treatment of post-inflammatory hyperpigmentation.

DETAILED DESCRIPTION:
Post-inflammatory hyperpigmentation is a common pigmentary skin disorder that is refractory to treatment and troublesome for darker skin individuals. The current treatment with conventional bleaching cream may result in skin irritation and ochronosis that is irreversible. Recent studies have shown that the topical cysteamine cream is safe and effective for dark spots such as melasma and lentigo with no significant side effects.

The primary aim of this study is to evaluate the safety and efficacy of topical cysteamine for postinflammatory hyperpigmentation. We conduct a randomized control, double-blinded trial to include 40 patients with postinflammatory hyperpigmentation. Clinical photography with VISIA skin imaging system,mexameter, transepidermal water loss, optical coherence tomography were used to evaluate the efficacy of treatment on a monthly basis for four months period. The patient was evaluated by two blinded investigator using the investigator global assessment. Patient global assessment was also recorded monthly.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* Patients with postinflammatory hyperpigmentation for more than 3 months.

Exclusion Criteria:

* Patients with topical hydroquinone, oral tranexamic acid and/or other skin whitening agents.
* Patients that receive or planning to receive laser treatment for spot removal during the study period.
* Individuals with allergic history to cysteamine or vehicle ingredients.
* Pregnant patients or patients planning to become pregnant during the time of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pigmentation at 4 Weeks | 4 weeks
  Patients will have their lesion pigmentation scored with the hyperpigmentation index after 4 weeks
Change from Baseline Pigmentation at 8 Weeks | 8 weeks
  Patients will have their lesion pigmentation scored with the hyperpigmentation index after 8 weeks
Change from Baseline Pigmentation at 12 Weeks | 12 weeks
  Patients will have their lesion pigmentation scored with the hyperpigmentation index after 12 weeks
Change from Baseline Pigmentation at 16 Weeks | 16 weeks
  Patients will have their lesion pigmentation scored with the hyperpigmentation index after 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ahramiyanpour N, Saki N, Akbari Z, Shamsi-Meymandi S, Amiri R, Heiran A. Efficacy of topical cysteamine hydrochloride in treating melasma: a systematic review. J Cosmet Dermatol. 2021 Nov;20(11):3593-3602. doi: 10.1111/jocd.14494. Epub 2021 Sep 30. PMID 34591360
- [Result] Nguyen J, Remyn L, Chung IY, Honigman A, Gourani-Tehrani S, Wutami I, Wong C, Paul E, Rodrigues M. Evaluation of the efficacy of cysteamine cream compared to hydroquinone in the treatment of melasma: A randomised, double-blinded trial. Australas J Dermatol. 2021 Feb;62(1):e41-e46. doi: 10.1111/ajd.13432. Epub 2020 Sep 27. PMID 32981068
- [Result] Karrabi M, David J, Sahebkar M. Clinical evaluation of efficacy, safety and tolerability of cysteamine 5% cream in comparison with modified Kligman's formula in subjects with epidermal melasma: A randomized, double-blind clinical trial study. Skin Res Technol. 2021 Jan;27(1):24-31. doi: 10.1111/srt.12901. Epub 2020 Jun 25. PMID 32585079
- [Result] Farshi S, Mansouri P, Kasraee B. Efficacy of cysteamine cream in the treatment of epidermal melasma, evaluating by Dermacatch as a new measurement method: a randomized double blind placebo controlled study. J Dermatolog Treat. 2018 Mar;29(2):182-189. doi: 10.1080/09546634.2017.1351608. Epub 2017 Jul 26. PMID 28678558
- [Result] Mansouri P, Farshi S, Hashemi Z, Kasraee B. Evaluation of the efficacy of cysteamine 5% cream in the treatment of epidermal melasma: a randomized double-blind placebo-controlled trial. Br J Dermatol. 2015 Jul;173(1):209-17. doi: 10.1111/bjd.13424. Epub 2015 May 29. PMID 25251767
- [Result] Karrabi M, Mansournia MA, Sharestanaki E, Abdollahnejad Y, Sahebkar M. Clinical evaluation of efficacy and tolerability of cysteamine 5% cream in comparison with tranexamic acid mesotherapy in subjects with melasma: a single-blind, randomized clinical trial study. Arch Dermatol Res. 2021 Sep;313(7):539-547. doi: 10.1007/s00403-020-02133-7. Epub 2020 Sep 2. PMID 32879998